CLINICAL TRIAL: NCT05996523
Title: Phase II Trial of Immunotherapeutic HPV Vaccine PRGN-2009 With Pembrolizumab Before Standard Treatment in Subjects With Newly Diagnosed HPV-Associated Oropharyngeal Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10001536; 001536-C
Record Dates: First submitted 2023-08-16; First posted 2023-08-18 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10-01

CONDITIONS: Oropharyngeal Squamous Cell Carcinoma (SCC)
Keywords: HPV16/18; PD-1 inhibitor; Monoclonal Antibody
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): PRGN 5x10^11 Viral Particles (VP) SC plus pembrolizumab 200mg IV as induction/ neoadjuvant therapy
  Interventions: Biological: PRGN-2009; Drug: Pembrolizumab

INTERVENTIONS:
Biological: PRGN-2009 — PRGN-2009 5x10^11 viral particles (VP) subcutaneously (SC) approximately two weeks apart
Drug: Pembrolizumab — Pembrolizumab 200 mg intravenously (IV) concurrently with the first vaccine dose

SUMMARY:
Background:

Cancers in and around the mouth associated with human papilloma virus (HPV) are common. Two treatments (the drug pembrolizumab and the HPV vaccine PRGN-2009) have been shown to work well when used individually against these cancers. Researchers want to find out if they might work better when used together.

Objective:

To test pembrolizumab combined with PRGN-2009 in people with HPV-positive cancers in and around the mouth.

Eligibility:

Adults aged 18 and older newly diagnosed with HPV-positive cancers in and around the mouth.

Design:

Participants will be screened. They will have a physical exam with blood tests. They will have imaging scans. They may need to have a biopsy: A sample of tissue will be taken from the tumor.

PRGN-2009 is given as an injection under the skin. Pembrolizumab is given through a tube attached to a needle inserted into a vein in the arm.

Participants will have at least 3 clinic visits: At the first, they will receive both the drug and the vaccine; 15 days later, they will receive a second shot of the vaccine. At the third visit, about 1 week after the second, they will have follow-up tests.

During these visits, participants will give samples of blood, urine, and saliva. Imaging scans and biopsies will be repeated. They will have tests of their heart function.

Participants may opt to return for another follow-up visit about 1 month after their second dose of the vaccine.

Participants will have follow-up contacts by phone 3 and 6 months after starting the study. The calls will continue once a year for 5 years.

DETAILED DESCRIPTION:
Background

-Human papilloma virus-associated oropharyngeal cancer (HPV-OPC) is the most common HPV-associated malignancy in the United States, with an increasing incidence. Although the prognosis for stage I HPV-OPC is favorable, about 20 percent of patients with stage II

disease and 35 percent of patients with stage III disease will die within four years.

* The standard-of-care primary treatment for HPV-OPC without distant metastasis is definitive concurrent chemoradiotherapy (primarily) or surgery (which may be followed by adjuvant chemoradiotherapy).
* Neoadjuvant/induction immunotherapy is in clinical trials aiming to induce antigen-specific immunity prior to primary treatment and to reduce the risk of disease relapse. Pembrolizumab, an anti-PD-1 monoclonal antibody that is FDA-approved for first-line treatment of recurrent/metastatic head and neck squamous cell cancer (HNSCC) has been used in these trials and shown to be safe and active.
* PRGN-2009 is an anti-HPV immunotherapeutic vaccine. It has demonstrated induction of HPV antigen-specific responses and tumor growth inhibition in pre-clinical models of HPV-associated malignancy, with improved anti-tumor efficacy upon addition of T-cell immune checkpoint blockade. In a Phase I/II trial at the NCI it has demonstrated excellent safety and tolerability as monotherapy or in combination with checkpoint blockade in recurrent/metastatic disease but also as monotherapy in neoadjuvant/induction context for HPV-OPC.

Objective:

-To determine if the use of PRGN-2009 with pembrolizumab in participants with p16-positive OPC can result in a >= 2-fold increase in CD3+ tumor infiltrating T cells post treatment compared with pre-treatment.

Eligibility:

* Age >= 18 years.
* Pathologically confirmed newly diagnosed Stage I (T1, T2; N1), II or III p16-positive OPC.

Design:

* This is a Phase II study to evaluate the effect of PRGN-2009 and pembrolizumab before definitive treatment in subjects with p16-positive OPC.
* Participants will receive PRGN-2009 and pembrolizumab prior to definitive treatment.
* Participants will receive two doses of PRGN-2009 5x10^11 viral particles (VP) subcutaneously (SC) approximately two weeks apart, and one dose of pembrolizumab 200 mg intravenously (IV) concurrently with the first vaccine dose.
* Up to 20 evaluable participants will be enrolled.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Subjects must have cytologically or histologically confirmed newly diagnosed stage I (T1,2 N1), II or III p16-positive oropharyngeal squamous cell carcinoma (SCC) planned for definitive therapy (surgery or chemoradiotherapy).
* Subjects must have measurable disease, per RECIST 1.1.
* Age >=18 years.
* Eastern Cooperative Oncology Group [ECOG] performance status <= 2.
* Adequate hematologic function at screening, as follows:

  * Absolute neutrophil count (ANC) >=1 x 10^9/L;
  * Hemoglobin (Hgb) >= 9 g/dL;
  * Platelets >= 75,000/microliter.
* Adequate renal and hepatic function at screening, as follows:

  * Serum creatinine <= 1.5 x upper limit of normal (ULN) OR measured or calculated creatinine clearance >= 40 mL/min for participant with creatinine levels > 1.5 x ULN (glomerular filtration rate [GFR] can also be used in place of creatinine or CrCl);
  * Total bilirubin <= 1.5 x ULN OR in subjects with Gilbert s syndrome, a total bilirubin <= 3.0 x ULN;
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <= 2.5 x ULN, unless liver metastases are present, then values must be <= 3 x ULN.
* Participants serologically positive for HIV, Hepatitis B, or Hepatitis C are eligible if the viral loads are undetectable by quantitative PCR. Note: HIV positive participants must have CD4 count >= 200 cells/mm^3 at enrollment, be on stable antiretroviral therapy for at least 4 weeks and have no reported opportunistic infections or Castleman s disease within 12 months prior to enrollment.
* Women of child-bearing potential (WOCBP) must agree to use effective contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and for at least 4 months following the last dose of pembrolizumab.
* Participants must be willing to undergo two research biopsies on this study.
* Ability of participant to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Participants with prior investigational drug, live vaccine, chemotherapy, immunotherapy, or any prior radiotherapy (except for palliative bone directed therapy) within the past 4 weeks prior to the first drug administration. Participants may continue adjuvant hormonal therapy in the setting of a definitively treated cancer (e.g., breast).
* Major surgery within 28 days prior to the first drug administration (minimally invasive procedures such as diagnostic biopsies are permitted).
* Pregnant individuals as evaluated by a positive serum or urine Beta-hCG at screening
* Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent with the exception of:

  * Diabetes type I, eczema, vitiligo, alopecia, psoriasis, hypo- or hyperthyroidism or other mild autoimmune disorders not requiring immunosuppressive treatment.
  * Administration of glucocorticoids through a route known to result in a minimal systemic exposure (topical, intranasal, intraocular, or inhalation).
* Systemic (intravenous or oral) glucocorticoid (except for physiologic doses of corticosteroids, i.e., <= the equivalent of prednisone 10 mg/day) or other immunosuppressors such as azathioprine or cyclosporin A, are excluded because of potential immune suppression. These treatments must be discontinued at least 1 week prior to enrollment for recent short course use (<= 14 days). Glucocorticoids as premedication for contrast-enhanced studies is allowed prior to enrollment and on study.
* Participants with a prior or concurrent malignancy whose natural history or treatment that has potential to interfere with the safety or efficacy assessment of the regimen.
* Prior allogenic tissue/solid organ transplant.
* Participants with pulse oximetry < 92% on room air at screening.
* Uncontrolled intercurrent illness that would limit compliance with study requirements suggested by medical history, physical examination or standard clinical assessments such as imaging and laboratory studies.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-11-07 (Actual); Primary Completion 2025-05-22 (Actual); Study Completion 2030-07-16 (Estimated)

PRIMARY OUTCOMES:
Determine if there is an increase in CD3+ tumor infiltrating T cells post treatment compared with pre-treatment | 4-5 weeks
  CD3+ tumor infiltrating lymphocytes will be assessed by multiplex immunofluorescence from the surgical/ biopsy tissue collected at week 4-5 and compared with pre-treatment

SECONDARY OUTCOMES:
Prolonged Survival | 3-6 months
  Assess if PRGN-2009 plus pembrolizumab results in significantly prolonged survival as compared to the expected 80% three-year historical survival in p16-positive OPC participants
Overall Survival | 5 years
  Assess OS and RFS once a year for 5 years
Safety | Up to 28 days after last treatment
  Incidence of treatment-related serious adverse events at baseline, W1, W3, on day 29, and 28 days after last treatment as defined by Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Determine the rate of increase in TILs by immunohistologyCHANGE TO: Determine the rate of increase in tumor infiltrating lymphocytes (TILs) by immunohistology | 4 weeks CHANGE TO: 4-5 weeks
  Compare the induction of immune response of PRGN-2009 plus pembrolizumab with PRGN-2009 at completion visit compared with pre-treatment with endpoint the >=2-fold increase in tumor infiltrating lymphocytes

CONTACTS AND LOCATIONS:
Overall Officials: Charalampos Floudas, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will be shared.@@@@@@All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.@@@@@@
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data from this study may be requested from other researchers no sooner than 3 years after the completion of the primary endpoint.@@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active@@@@@@@@@@@@
Access Criteria: Data from this study may be requested by contacting the PI@@@@@@Genomic data are made available via dbGaP through requests to the data custodians.@@@@@@

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_001536-C.html